CLINICAL TRIAL: NCT07363681
Title: Beyond Inhalational Agents: Dexmedetomidine for Maintenance of General Anesthesia - A Prospective Randomized Clinical Trial
Brief Title: Inhalational Agents Versus Dexmedetomidine for Maintenance of General Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Nalan Saygi Emir, Specialist Physician, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/176
Record Dates: First submitted 2025-12-17; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-06

CONDITIONS: Ureterorenoscopic Lithotripsy; Transurethral Resection of the Bladder; Percutaneous Nephrolithotomy; Transurethral Resection of the Prostate
MeSH Terms: interventions — Dexmedetomidine; Remifentanil; Desflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group DR: Dexmedetomidine + Remifentanil (Active Comparator): The investigators will administer dexmedetomidine combined with remifentanil for anesthesia maintenance in this patient group.
  Interventions: Drug: Dexmedetomidine + Remifentanil
- Group IR: Desflurane + Remifentanil (Active Comparator): The investigators will administer desflurane combined with remifentanil for general anesthesia maintenance in this group.
  Interventions: Drug: Desflurane + Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine + Remifentanil — Anesthesia Protocol
  All patients will receive the same standardized induction regimen consisting of fentanyl (1 μg/kg), propofol (1 mg/kg), and rocuronium (0.5 mg/kg). Following induction, maintenance of general anesthesia will differ according to group allocation:
  In Group DR, anesthesia maintenance will be provided with dexmedetomidine administered as a continuous infusion without a loading dose, combined with remifentanil infusion.
  Remifentanil infusion rates will be adjusted as clinically required to maintain adequate hemodynamic stability and surgical anesthesia depth
  Arms: Group DR: Dexmedetomidine + Remifentanil
Drug: Desflurane + Remifentanil — The investigators will administer desflurane combined with remifentanil for general anesthesia maintenance in this group.
  Arms: Group IR: Desflurane + Remifentanil

SUMMARY:
The climate crisis and environmental pollution are escalating day by day, making the reduction of carbon footprints increasingly important both on an individual and industrial level. Inhalational anesthetic agents are widely used in daily anesthesia practice. However, some of these agents are released into the environment either unchanged or as metabolic by-products. It can take hundreds of years for these substances to be fully eliminated from nature. Therefore, there is a growing interest in identifying alternative anesthetic agents that are fully metabolized, do not produce waste, have a shorter duration of action, and pose less harm to ecosystems.

Recent clinical studies have shown that dexmedetomidine, when administered intraoperatively via infusion without a loading dose and in combination with inhalational agents, provides more stable hemodynamics and results in a shorter postoperative recovery period. Commonly used as a long-term sedative agent in intensive care units, dexmedetomidine has gained popularity in the intraoperative setting due to its stable hemodynamic profile, low incidence of withdrawal symptoms, and faster recovery.

In this study, it is aimed to demonstrate the potential use of dexmedetomidine-whose pharmacodynamic and pharmacokinetic properties are well-known to experienced anesthesiologists-as an alternative to inhalational anesthetic agents for the maintenance of anesthesia, particularly in the geriatric patient population.

DETAILED DESCRIPTION:
Study Design and Setting This prospective, randomized clinical study was conducted at the Department of Anesthesiology and Reanimation, University of Health Sciences, Bakırköy Dr. Sadi Konuk Training and Research Hospital. Patient randomization was performed using a computer-based randomization tool (@randomizer).

Patient Selection A total of 150 patients over the age of 39 who provided informed consent and were scheduled for elective urological procedures at the Urology Department were enrolled in the study. The included surgeries were uretero-renoscopic lithotripsy (URS), transurethral resection of the bladder (TUR-B), percutaneous nephrolithotomy (PCNL), and transurethral resection of the prostate (TUR-P).

Anesthesia Protocol

Upon arrival to the operating room, standard monitoring was applied to all patients. Anesthesia induction and maintenance were carried out according to randomization:

Group DR: Dexmedetomidine + Remifentanil

Group IR: Desflurane + Remifentanil

Intraoperative and Postoperative Data Collection

During surgery, anesthesia depth and hemodynamic parameters were continuously monitored and recorded. At the end of the procedure, the following postoperative data were collected:

Visual Analog Scale (VAS) for pain

Richmond Agitation-Sedation Scale (RASS)

Modified Aldrete Score

The hospital unit/ward to which the patient was transferred

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 39 years
* Classified as ASA physical status II-IV
* Scheduled for elective endoscopic urological surgery (e.g., URS, TUR-B, PCNL, TUR-P)
* Scheduled for postoperative follow-up in the Post-Anesthesia Care Unit (PACU)
* Ability to provide written informed consent

Exclusion Criteria

* Requirement for conversion to open surgery during the perioperative period
* Patients who decline to participate in the study
* Presence of neuropsychiatric disorders (e.g., dementia, Parkinson's disease, epilepsy, or history of head trauma)
* History of alcohol or substance abuse
* Use of psychoactive medications
* Inability to communicate adequately for any reason

Ages: 39 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
Depth of anesthesia | Intraoperative period
  Depth of anesthesia assessed using Bispectral Index (BIS) monitoring, with BIS values recorded during surgery. The target BIS range will be 40-60.

SECONDARY OUTCOMES:
Intraoperative hemodynamic stability | Intraoperative period
  Intraoperative hemodynamic stability assessed by mean arterial pressure (MAP) and heart rate (HR) values recorded during surgery.
Quality of recovery | Postoperative day 1
  Quality of recovery assessed using the Quality of Recovery-15 (QoR-15) questionnaire (score range 0-150; higher scores indicate better recovery).
Sedation Level | Post-anesthesia care unit (PACU)
  Sedation level assessed using the Richmond Agitation-Sedation Scale (RASS) (score range -5 to +4) where more negative scores indicate deeper sedation and positive scores indicate agitation

OTHER OUTCOMES:
Postoperative recovery time | Post-anesthesia care unit (PACU)
  Postoperative recovery time defined as the time to achieve an Aldrete score ≥9.
Postoperative pain intensity | Up to 24 hours postoperatively
  Postoperative pain intensity assessed using the Visual Analog Scale (VAS; 0-10), where higher scores indicate worse pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy dr. Sadi Konuk, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF